CLINICAL TRIAL: NCT02381002
Title: EVALUATION OF DIETARY REGIMEN AND PHYSICAL ACTIVITY ON IRON AND LIPID STATUS IN OVERWEIGHT AND OBESE CHILDREN 6 Months Prospective Study
Brief Title: Effect of Weight Reduction Program on Overweight and Obese Children
Acronym: "ironobese"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics , Faculty of Medicine, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FMASU 1078/2012
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Childhood Obesity
Keywords: Serum ferritin, physical exercise, Diet
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weight reduction (Experimental): weight reduction program for 6 months
  Interventions: Other: Weight reduction program

INTERVENTIONS:
Other: Weight reduction program — Overweight and obese children (6-12 years old) from patient group accepting enrollment were assigned to weight reduction program for 6 months with monthly follow up. The program comprise: 1) Diet regimen: Healthy balanced diet was prescribed. The amount of calories was determined according to 24-hour recall then 250-500 calories were subtracted from total intake which decrease weight by 0.25-0.5 kg/week. 2) Exercise:were instructed to practice walking for at least 30 minutes 3-4 times per week.

SUMMARY:
Background: Obesity is associated with alterations in iron metabolism leading to iron deficiency.

Aim: to study the prevalence of obesity among primary school students, assess iron status among overweight/obese children with age ranging between 6 and 12 years and the effect of weight reduction program on iron status.

Patients and Methods: The study will be conducted on 2 groups. Group 1 will include 1025 primary school children recruited from 2 urban schools in Cairo with age ranging between 6 and 12. Anthropometric measures and prevalence of overweight/obesity will be assessed. Group 2 will include 100 obese children according to the CDC definition and 50 age and sex matched children with normal weight. All will be subjected to history taking, anthropometric measures, complete blood picture, iron profile and soluble transferrin receptor. Weight reduction program for 6 months will be done for obese children and all parameters will be re-ckecked.

DETAILED DESCRIPTION:
SUMMARY Over the past 30 years, childhood overweight/obesity, often beginning in infancy and toddlerhood, has reached epidemic proportions, particularly among minority and/or low-income populations in high-income countries. Rates of pediatric obesity (BMI ≥ 95th percentile) have almost tripled over the past 25 years, with current estimates showing a prevalence rate of 16% for girls and 18% for boys. The prevalence of adolescent and childhood overweight and obesity in children living in Egypt, Brazil and Mexico has reached levels comparable to those seen in industrialized nations.

Obesity is associated with alterations in iron metabolism leading to iron deficiency which is probably the most prevalent single common micronutrient deficiency in the world today.

Aim of the study :

1. To assess iron status among overweight/ obese primary school children. With age ranging from 6 years till preadolescence or age 12 years with Tanner score ≤ 2.
2. To assess the effect of 6 months dieting program on iron status improvement in overweight/obese children.
3. To study the psychological basis of obesity in children as well as associated co-morbidities.
4. To assess the prevalence of obesity among primary school students.

The study will be conducted on 2 groups:

Group 1 1025 will be recruited from 2 urban primary schools with moderate-high social standards among children with age between 6 to 12 years.

Weight, height were measured and body mass index will be calculated. All measures will be plotted on the percentiles for age. The percentage of obese and overweight children will be calculated.

Group 2 will include 150 children, 100 obese children and 50 normal weight children with age ranging between 6 and 12 years.

All 150 subjects will be subjected to:

1. A questionnaire: inquiring about personal data, Socioeconomic data, family history of obesity, weight related attitudes, physical exercise performance, personal believes about diet (self-efficacy, barriers to change and dietary believes), previous trials to lose weight and school performance.
2. Full clinical examination: including

   1. Systemic examination and blood pressure measurements.
   2. Anthropometric measurements which include weight, height and body mass index.
3. Laboratory investigations: complete blood picture, serum iron, ferritin, transferrin saturation, total iron binding capacity, soluble transferrin receptor, serum triglycerides and serum cholesterol.

All obese children will be subjected to weight reduction program which includes diet regimen, exercise and behavioral modification.

All anthropometric and laboratory measures will be measured again after the 6 months intervention.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese children according to BMI percentiles with age between 6 and 12 years.

Exclusion Criteria:

* Obesity caused by genetic syndromes, apparent endocrinal disease, psychiatric disorders or chronic inflammatory diseases (inflammatory bowel disease, autoimmune disease, cancer treated within the last year).
* Children with chronic illness or blood disorders such as any identified risk for iron deficiency or a red cell disorder, vegan diet.
* Children with Tanner>2

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Successful weight reduction (>5% weight loss at 6 months). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S Elalfy, PhD, MD, Study Chair — Pediatric department, Faculty of Medicine , Ain Shams University
Locations (1):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt